CLINICAL TRIAL: NCT04481841
Title: Head Yuanshi Dian Therapy in the Treatment of Burning Mouth Syndrome: a Randomized Controlled Trial
Brief Title: Head Yuanshi Dian Therapy in Burning Mouth Syndrome
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang Provincial Hospital of TCM (Other); Guiyang Hospital of Stomatology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-281
Record Dates: First submitted 2019-11-15; First posted 2020-07-22 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-01

CONDITIONS: Burning Mouth Syndrome; Oral Mucosa Disease
Keywords: Burning Mouth Syndrome; Effect and Safety; Primary Point Push
MeSH Terms: conditions — Burning Mouth Syndrome | interventions — gamma-oryzanol; Riboflavin; Vitamin E

STUDY DESIGN:
Intervention Model Description: 1:1 randomized controlled clinical trial were used. Random numbers generated by SPSS21.0 will be placed in sequentially coded, sealed, opaque envelopes. When the qualifications of the subjects were determined by the researchers, the envelopes were opened sequentially and the subjects were assigned to groups. The odd number represented the experimental group and the even number represented the control group.
Who Masked: Outcomes Assessor
Masking Description: Each of the three centers has a researcher responsible for the treatment and interpretation of the subjects. The head of the research center trained the researcher to unify the standards. Three researchers were not involved in the evaluation of efficacy. Another researcher was responsible for recording pain and emotional nature and degree score, pain index, pain multi-dimensional characteristics score, depression index, Pittsburgh sleep quality index, Kupperman menopause score, dry mouth subjective symptoms questionnaire, saliva flow, and recording laboratory results, and collecting records. Data, analysis of efficacy, the researchers do not know the specific grouping, in order to minimize the subjective impact of the researchers on the test results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): On the basis of classical "Gu-Nucleus-E" triple drug therapy, the experimental group was treated with head yuanshi dian therapy twice a day for 1 months as a course of treatment.
  Interventions: Drug: oryzanol + vitamin B2 (riboflavin) + vitamin E
- control group (Active Comparator): oryzanol + vitamin B2 (riboflavin) + vitamin E, oryzanol tablets, oral, 10 mg/time, 3 times/day; vitamin B2 tablets, oral, 10 mg/time, 3 times/day; vitamin E pills, oral, 100 mg/time, 1 time/day, 1 months as a course of treatment.
  Interventions: Drug: oryzanol + vitamin B2 (riboflavin) + vitamin E

INTERVENTIONS:
Drug: oryzanol + vitamin B2 (riboflavin) + vitamin E — 1:Control group Specific medicines and usage, course of treatment are as follows: oryzanol + vitamin B2 (riboflavin) + vitamin E, oryzanol tablets, oral, 10 mg/time, 3 times/day; vitamin B2 tablets, oral, 10 mg/time, 3 times/day; vitamin E pills, oral, 100 mg/time, 1 time/day, 1 months as a course of treatment.
  2.Therapeutic regimen of experimental group On the basis of classical "Gu-Nucleus-E" triple drug therapy, the experimental group was treated with head yuanshi dian therapy twice a day for 1 months as a course of treatment.
  Other Names: head yuanshi dian therapy

SUMMARY:
Burning mouth syndrome is one of the most common oral mucosal diseases in clinic. It is a chronic pain syndrome with extensive burning pain of oral mucosa as its main symptoms. There are no pathological changes in oral mucosa and no characteristic histopathological changes. Patients often have accompanying symptoms such as depression and xerostomia. Although the patient does not have obvious oral lesions, the pain symptoms are more serious and the mental pressure is greater.

BMS, as a complex clinical syndrome associated with multiple factors, mainly occurs in people aged 27-87, with an average age of 61. BMS is rare among people under 30 years old. BMS is predominant in women, the ratio of male to female is 1:5 to 1:7, the incidence is 0.7%-15%, and increases with age. Up to 90% of female patients are in perimenopausal period. Symptoms occur from 3 years before menopause to 12 years after menopause.

The causes of BMS are complex, and the treatment is difficult, easy to relapse and protracted. Studies have confirmed that the occurrence and development of BMS are directly related to mental factors. Therefore, psychosocial factors are the most important pathogenic factors of BMS. If we intervene in these factors, it is hopeful to improve the curative effect of BMS.

Traditional psychotherapy methods include drug treatment, psychotherapy, surgical treatment, traditional Chinese medicine treatment, etc. Drug treatment is mainly based on different types of mental and psychological diseases, choose different pharmacological effects of drugs, so as to effectively control the disease. However, these drugs are prone to adverse reactions such as sleepiness, weight gain, headache, physical weakness, etc. The basic principle of psychotherapy is to let patients fully expose symptoms, listen to their complaints patiently, carry out explanatory psychotherapy according to their medical history or take other psychological training, so as to relieve patients' mental stress and alleviate symptoms. But this method has a long course of treatment and needs the cooperation of the patients' family members; the basic principle of surgical treatment is to resect the corresponding areas of the brain or adopt endoscopy and micro-current to treat them, but the risks and injuries caused by the operation are greater, and the adverse reactions after the operation are larger; the treatment of traditional Chinese medicine needs a long course of treatment, and the treatment of some patients. The effect is not stable enough.

The causes of BMS are complex, there is no objective disease in clinic, and the patients suffer from abnormal pain, but the treatment methods are not uniform, and the curative effect is not good, which makes the patients unable to get effective treatment in the early stage of the disease, and easy to relapse, resulting in the aggravation and development of BMS into intractable sensory abnormalities, and protracted! Literature reports confirm that the tri-drug of oryzanol-riboflavin-vitamin E (oryzanol-riboflavin-vitamin E) is a classic treatment for BMS and has been included in the classic book in China, Pharmacotherapy for oral mucosal disease . However, its long-term clinical application has found that its efficacy is unstable, and clinical symptoms after drug withdrawal. The symptoms are prone to recurrence or even aggravation. Therefore, it is necessary to use the classical program on the basis of a combination of interventions to promote the efficacy of stable and safe.

Over the past two years, the investigators has treated nearly 100 cases of BMS with head yuanshi dian therapy, and achieved satisfactory results. It can obviously relieve burning pain of BMS oral mucosa, promote saliva secretion, improve dry mouth and bitter mouth, and improve sleep to a certain extent. However, due to the limited number of cases treated, the classification of BMS is not meticulous enough, and there are still vague areas in the classification of BMS, which affects the rigorous evaluation of the therapeutic effect of BMS.

Therefore, the investigators propose a hypothesis: can the head yuanshi dian therapy be used as the main adjuvant therapy for BMS? By consulting Pubmed, OVID, CNKI, Wanfang and other major databases at home and abroad, the investigators found that there is no relevant report at home and abroad. In view of this, the investigators intend to design this randomized positive controlled clinical trial, using conventional valley-nucleus-E triple drug therapy as the positive control group, to observe the efficacy and safety of head yuanshi dian therapy for BMS, in order to find a safe and effective green non-invasive therapy, effectively alleviate or eliminate oral mucosal pain, dry mouth, etc.

DETAILED DESCRIPTION:
2.1 Test Target

To observe the efficacy and safety of head yuanshi dian therapy in the treatment of BMS.

2.2 Case Collection 2.2.1 Diagnostic criteria

1. Burning-like neuropathic pain occurs in the tongue or other parts of oral mucosa, which may be relieved or disappeared when attention is transferred.
2. Most of them are accompanied by dry mouth, numbness, taste disorder, depression, insomnia and other emotional changes, neuropathological changes;
3. Symptom changes may have special regularities and rhythms, such as mild morning symptoms and worsening afternoon symptoms; pain does not increase when eating or drinking water, and usually does not affect sleep; or persistent pain; or intermittent throughout the day;

2.2.3 Exclusion criteria

1. There are local stimulating factors that can cause burning pain in the mouth (including bad prosthesis, sharp cusp or ridge, complete denture, etc.).
2. Patients with other serious oral mucosal diseases (including bullous diseases, allergic diseases, oral candidiasis, oral lichen planus, recurrent aphthous ulcer, etc.);

2.2.4 Standards and procedures for discontinuation of trial/trial therapy When the following occurs, the trial can be stopped according to the judgement of the researcher, and the reasons for the discontinuation of the trial can be recorded in the case report form (CRF) and the original record. If the cause of adverse events leads to the discontinuation of the test, the relevant treatment should be carried out according to the adverse events.

1. Misacceptance was found after enrollment;
2. Those who received neurological, psychiatric drugs or other interventions during the trial;
3. Those who did not use the test drug according to the doctor's advice or who were treated by the combination of internal and external heat source and push of the original point after admission into the group;

2.3 randomization In this study, multi-center (Zhejiang University Second Hospital, Zhejiang Hospital of Traditional Chinese Medicine, Guiyang Hospital of Stomatology, Guizhou, 3 clinical research centers), non-inferior effect, 1:1 randomized controlled clinical trial were used. Random numbers generated by SPSS21.0 will be placed in sequentially coded, sealed, opaque envelopes. When the qualifications of the subjects were determined by the researchers, the envelopes were opened sequentially and the subjects were assigned to groups. The odd number represented the experimental group and the even number represented the control group.

2.4 Measures to Reduce and Avoid Bias In order to reduce and avoid the bias of experimental conditions, the investigators should strictly group according to the random number of groups, and adopt the corresponding treatment plan. At the same time, in order to ensure the objectivity of the study group's evaluation of cases dropped and excluded, it is necessary to clarify the statistical treatment methods and evaluation criteria for cases dropped and excluded in the statistical analysis plan.

2.5 Sample size calculation Referring to the previous study of this group, the difference and standard deviation of the mean between the two groups before treatment and after one month of treatment were used to calculate the sample size required for this study. Based on the visual analogue scale (VAS), the non-inferior boundary value was allowed to be 1 and the standard deviation was 2.3, and 113 persons were needed for each group (90% of the test efficiency and 0.025 of the alpha). Taking into account the possibility of abscission, 290 cases were finally included.

2.6 Researcher and patient training The main researcher receives relevant training in head yuanshi dian therapy, and can master the principle of the therapy and related matters needing attention, as well as the use of various psychological dosimeters. In addition, the main researcher trained the patients in this therapy so that they could take care of themselves at home.

2.7 Basic information of subjects During the first and second visits, the investigators recorded the basic information of the subjects in the BMS Case Report Form: case number, random number, visiting date, name, sex, age, occupation, employment status, education level, contact mode, nationality, communication address, systemic disease, allergy history, medication history, and so on. Family history, female subjects recorded menstrual history, routine physical examination results, etc.

2.8 Trial Groups and Treatment Programs 2.8.1 Treatment plan of control group Specific medicines and usage, course of treatment are as follows: oryzanol + vitamin B2 (riboflavin) + vitamin E, oryzanol tablets, oral, 10 mg/time, 3 times/day; vitamin B2 tablets, oral, 10 mg/time, 3 times/day; vitamin E pills, oral, 100 mg/time, 1 time/day, 1 months as a course of treatment.

2.8.2 Therapeutic regimen of experimental group On the basis of classical "Gu-Nucleus-E" triple drug therapy, the experimental group was treated with head yuanshi dian therapy twice a day for 1 months as a course of treatment.

2.8.3 Specific operating procedure of head yuanshi dian therapy

2.9 Evaluation Index of Therapeutic Effect After the first visit or passing the push maneuver retraining, participants will have a visit twice a week. The aim is to observe the efficacy and safety of the treatment. At the end of one week, two weeks, three weeks and one month of treatment, the researchers recorded the efficacy indicators of the patients. The immunoglobulin, hemorheology index, blood routine, ESR, CRP, blood lipid routine and changes were examined at the first diagnosis and at the end of treatment. At the end of the treatment, the drug was stopped, and the head Yuanshi Dian therapy was suspended in the experimental group. The patients were followed up one month after the treatment and three or six months after the treatment by telephone to observe the recurrence.

2.10 Blind Assessment Each of the three centers has a researcher responsible for the treatment and interpretation of the subjects. The head of the research center trained the researcher to unify the standards. Three researchers were not involved in the evaluation of efficacy. Another researcher was responsible for recording pain and emotional nature and degree score, pain index, pain multi-dimensional characteristics score, depression index, Pittsburgh sleep quality index, Kupperman menopause score, dry mouth subjective symptoms questionnaire, saliva flow, and recording laboratory results, and collecting records. Data, analysis of efficacy, the researchers do not know the specific grouping, in order to minimize the subjective impact of the researchers on the test results.

2.11 Safety Evaluation Index 2.11.1 Laboratory Indicators Two groups of subjects were required to provide the following examination reports within 12 months: blood routine, blood sugar, liver and kidney function, urine routine, abdominal ultrasonography, chest X-ray, sex hormone levels.

2.11.2 Indicators of vital signs Including blood pressure and pulse. 2.11.3 Adverse reactions The subjects in the experimental group can inform the researchers of any discomfort and have the right to withdraw from the trial at any time when they are given the head yuanshi dian therapy. When the subjects in the control group were re-visited, the researchers asked if there were any adverse reactions during the medication process. If so, they should record in detail, including the number of adverse reactions (incidence), specific reactions, elimination and so on.

ELIGIBILITY:
Inclusion Criteria:

* Persons aged 25-90;
* By inquiring the medical history in detail, BMS can be diagnosed if the clinical symptoms and signs do not conform to the clinical characteristics, and the medical history is more than 4 months.
* Burning pain and/or dry mouth in tongue or other parts of oral mucosa were the main clinical symptoms.
* Those with normal blood routine, blood sugar, liver and kidney function, urine routine, abdominal ultrasonography, chest X-ray and other basic physical examination items;
* Those who voluntarily participate in the experiment and sign the informed consent.

Exclusion Criteria:

* There are local stimulating factors that can cause burning pain in the mouth;
* Patients with other serious oral mucosal diseases;
* Complicated with serious systemic diseases;
* Patients with mental disorders who take drugs routinely;
* Abnormal levels of sex hormones;
* Sjogren's syndrome.
* Possible drug-related xerostomia.
* Pregnant or lactating women;
* The patients'cognitive level was low and they could not understand and fill in the questionnaire correctly.
* Those who fail to comply with the doctor's advice or return to the doctor on time;
* Those who participated in clinical trials within 3 months.

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2020-07-27 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain index | one year
  The basic method is to use a swimming scale about 10 cm long, with 10 scales on one side, and the two ends are "0" and "10" ends respectively. 0 indicates no pain and 10 points represents the most severe pain that is unbearable.
Depressive mood index | one year
Pittsburgh sleep quality index | one year
Kupperman Climacteric Score | one year

CONTACTS AND LOCATIONS:
Overall Officials: Weilian Sun, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (3):
- China (3):
  - Guiyang Hospital of Stomatology, Guiyang, Guizhou
  - Zhejiang Provincal Hospital of TCM, Hangzhou, Zhejiang
  - Department of Oral Medicine, the Second Affiliated Hospital, School of Medicine Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No